CLINICAL TRIAL: NCT06969274
Title: Ultrasound-guided Sacral Erector Spinae Plane Block as a Sole Anesthetic Technique Versus Saddle Block in Hemorrhoidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer of anesthesia, intensive care and pain medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAMSU R83/2025
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SESPB (Experimental)
  Interventions: Procedure: Ultrasound guided sacral erector spinae plane block (SESPB)
- Saddle (Experimental)
  Interventions: Procedure: Saddle block.

INTERVENTIONS:
Procedure: Ultrasound guided sacral erector spinae plane block (SESPB) — Patients will receive an Ultrasound guided sacral erector spinae plane block (SESPB)
  Arms: SESPB
Procedure: Saddle block. — Patients will receive a Saddle block.
  Arms: Saddle

SUMMARY:
Study interventions:

The patients will be randomized into two equal groups, Group A and Group B.

Group A: Patients will receive an Ultrasound guided sacral erector spinae plane block (SESPB)

Group B: Patients will receive Saddle block.

The surgical procedure will be performed by an experienced surgeon.

The outcome:

The primary outcome will be assessment of pain intensity using the NRS ranging from 0 (no pain) to 10 (worst pain) at 0, 2, 4, 6, 12, and 24 hours after the procedure. The secondary outcomes will include the cumulative doses of tramadol (50 mg intramuscular) to be repeated every 8 hours in case NRS score is more than four, the number of patients requiring rescue medication in the postoperative period.

DETAILED DESCRIPTION:
Study interventions:

The patients will be randomized into two equal groups using a computer-generated random numbers table, named Group A and Group B. An independent data manager, utilizing computer generated software, will be responsible for the randomization process. Patients will be assigned to the groups through sequentially numbered, sealed, opaque envelopes containing the computer-generated random numbers, which will be accessible only to the anesthesiologist performing the block. The subjects will be randomly allocated to one of the two groups.

Group A: Patients will receive an Ultrasound guided sacral erector spinae plane block (SESPB)

Group B: Patients will receive Saddle block.

Preoperatively, history taking, clinical examination and routine laboratory investigation will be performed, patients will be instructed to fast for 6 hours for solids and 2 hours for clear fluids. Upon arrival in the operation room, intravenous access will be established, and an acetated ringer's solution will be infused at a rate of 10ml/kg. ECG, noninvasive blood pressure and arterial oxygen saturation will be routinely monitored. The Numerical Rating Scale (NRS) will be used to assess pain intensity, and all study participants will be trained preoperatively to use the NRS pain score system.

In the operating room, a 20 G peripheral intravenous (IV) cannula will be inserted. Baseline parameters including a five-lead electrocardiogram (ECG), non-invasive blood pressure and peripheral oxygen saturation will be recorded. Intravenous midazolam at a dose of 0.02 mg/kg will then be administered.

The procedure in both groups will be performed by Dr. Riham Fathy Galal who is an anesthesiology consultant.

In group A, following asepsis protocols, patients will undergo a procedure in which a linear ultrasound probe (10-15 MHz)-Sono site M-turbo ultrasonography will be positioned on the transverse plane, specifically on the fifth spinous process. The probe will then be moved downward to visualize the first and second median sacral crests. Subsequently, the transducer will be placed 3 to 4 cm laterally to the second medial sacral crest to visualize the intermediate sacral crest. In the interfacial plane, 20 mL of local anesthetic solution (consisting of 10 mL of 0.5% bupivacaine, 5 mL of 2% lidocaine, and 5 mL of normal saline) will be injected using a 9-cm 22-gauge spinal needle between the erector spinae muscles and the intermediate sacral crest. The same procedure will be performed on the contralateral side.

In group B, Spinal anesthesia will be uniformly administered to the patient in the sitting position. A 25-gauge spinal needle (KDF, China) will be used to perform the spinal anesthesia at the L3-L4 or L4-L5 interspace. After confirming the presence of cerebrospinal fluid, 2 to 2.5 mL of 0.5% hyperbaric bupivacaine hydrochloride will be injected into the intrathecal space. The patients will then be placed in supine position.

After waiting 5 to 10 minutes to confirm that the spinal block level has reached the T10 dermatome, the patients will be repositioned into the lithotomy position. Oxygen will be administered via the nasal cannula at a rate of 2 L/min. If a decrease in blood pressure of greater than 20% from the baseline value is observed, ephedrine (0.1 mg/kg) will be administered. If the heart rate falls below 50 bpm, atropine (0.5 mg/ kg) will be administered.

An experienced surgeon will perform the surgical procedure. At the end of the operation, each patient will receive a single intravenous dose of paracetamol at 15 mg/kg, along with intravenous diclofenac at 1.5 mg/kg (with a maximum dose of 75 mg). During the postoperative period, all patients will receive intravenous paracetamol every 8 hours at a dose of 15 mg/kg, and intravenous diclofenac every 12 hours at a dose of 1.5 mg/kg (with a maximum dose of 75 mg). If the Numeric Rating Scale (NRS)score exceeded three, intravenous tramadol at a dose of 1.5 mg/kg will be administered as rescue analgesia.

The outcome:

The primary outcome will be assessment of pain intensity using the NRS ranging from 0 (no pain) to 10 (worst pain) at 0, 2, 4, 6, 12, and 24 hours after the procedure. The secondary outcomes will include the cumulative doses of tramadol (50 mg intramuscular) to be repeated every 8 hours in case NRS score is more than 4, the number of patients requiring rescue medication in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 18 to 65 years.
3. Both sexes.
4. Patients scheduled for perianal surgeries (hemorrhoidectomy).

Exclusion Criteria:

* 1- Patients with spinal malformation. 2-Patients with liver impairment. 3- Patients with renal impairment. 4-Patients younger than 18 years or older than 65 years. 5- Patients with hypersensitivity to one of the used drugs. 6- Coagulopathy disorders. 7- Patients who underwent hemorrhoidectomy before.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be assessment of pain intensity using the NRS ranging from 0 (no pain) to 10 (worst pain) at 12 hours after the procedure. | Twenty Four hours after the procedure
  The primary outcome will be assessment of pain intensity using the NRS ranging from 0 (no pain) to 10 (worst pain) at 12 hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No